CLINICAL TRIAL: NCT00538473
Title: Reactogenicity and Immunogenicity of GSK Biologicals' Influenza Vaccine GSK576389A in Elderly Adults (≥67 Years) Previously Vaccinated With the Same Candidate Vaccine. Fluarix™ Will be Used as Reference.
Brief Title: Evaluate Safety and Immunogenicity of GSK Bio's Influenza Vaccine GSK576389A After Repeated Vaccination in Elderly Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110223
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK576389A; Influenza Infection; Fluarix
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- FluAS25 (GSK576389A) Group (Experimental): Subjects received 1 dose of GlaxoSmithKline (GSK) Biologicals' AS25 adjuvanted influenza vaccine (GSK576389A).
  Interventions: Biological: GSK Biologicals' influenza vaccine GSK576389A
- Fluarix Group (Active Comparator): Subjects received 1 dose of Fluarix™.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: GSK Biologicals' influenza vaccine GSK576389A — Single dose, intramuscular injection
  Arms: FluAS25 (GSK576389A) Group
Biological: Fluarix™ — Single dose, intramuscular injection
  Arms: Fluarix Group

SUMMARY:
Since influenza vaccines are administered every year because of the frequent change in their antigenic composition, the safety and immunogenicity profile of GSK Biologicals' influenza vaccine GSK576389A will be re-evaluated after repeated vaccine administration. In this study, the subjects previously enrolled in study 107973 will receive a dose with the 2007-2008 season's formulations of Fluarix or GSK576389A. Only subjects who were previously enrolled in study 107973 (NCT00386113) are eligible for participation in this study.

DETAILED DESCRIPTION:
This study is a year 3 revaccination study. Second year revaccination was done in study 107973 (NCT00386113). First year revaccination was done in study 104540 (NCT00318058). Primary study was study 103304.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously vaccinated with GlaxoSmithKline Biologicals Fluarix™ or GSK576389A vaccines in the 107973 study (NCT00386113).
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged >= 67 years at the time of re-vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation (medical history and medical history directed examination) before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol up to 21 days after vaccination.
* Confirmed influenza infection since the date of previous vaccination.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Vaccination against influenza since January 2007 with the Northern Hemisphere 2007/2008 influenza vaccine or 2006/2007 influenza vaccine.
* Administration of more than 14 days of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s).
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation (medical history and medical history directed physical examination) or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which intramuscular injections are contraindicated.

Min Age: 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-10-23; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Started | 33 | 35
Completed | 32 | 35
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (4.53) | 73.2 (5.34) | 73.15 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include ecchymosis, pain, redness and swelling. Any: any symptom regardless of intensity grade. Grade 3 pain: considerable pain at rest, which prevented normal everyday activities. Grade 3 ecchymosis, redness and swelling: more than 100 millimeter.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 33 | 35
Subjects
  Any ecchymosis | 0 | 1
  Grade 3 ecchymosis | 0 | 0
  Any pain | 17 | 7
  Grade 3 pain | 0 | 0
  Any redness | 10 | 4
  Grade 3 redness | 1 | 0
  Any swelling | 2 | 2
  Grade 3 swelling | 0 | 0

2. Primary Outcome: Duration of Solicited Local Symptoms
Description: Duration was expressed as median number of days any symptom persisted. Solicited local symptoms assessed include ecchymosis, pain, redness and swelling. Any: occurrence of any local symptom regardless of their intensity grade.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on those subjects who reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 17 | 7
Days
  Ecchymosis (N= 0; 1) | NA [NA to NA] — No subjects experienced this symptom | 5.0 [5.0 to 5.0]
  Pain (N= 17; 7) | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Redness (N= 10; 4) | 2.5 [1.0 to 6.0] | 2.0 [1.0 to 2.0]
  Swelling (N= 2; 2) | 1.5 [1.0 to 2.0] | 2.5 [2.0 to 3.0]

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any: any symptom regardless of intensity grade; any fever: oral temperature greater than or equal to 38 degrees Celsius (°C). Grade 3: symptoms that prevented normal activity ; Grade 3 fever: oral temperature greater than 39°C. Related: symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 33 | 35
Subjects
  Any arthralgia | 8 | 5
  Grade 3 arthralgia | 0 | 0
  Related arthralgia | 7 | 1
  Any fatigue | 8 | 3
  Grade 3 fatigue | 0 | 0
  Related fatigue | 8 | 2
  Any headache | 8 | 3
  Grade 3 headache | 0 | 0
  Related headache | 6 | 2
  Any myalgia | 8 | 1
  Grade 3 myalgia | 0 | 0
  Related myalgia | 8 | 0
  Any nausea | 3 | 1
  Grade 3 nausea | 0 | 0
  Related nausea | 2 | 0
  Any shivering | 6 | 3
  Grade 3 shivering | 0 | 0
  Related shivering | 5 | 2
  Any fever | 1 | 0
  Grade 3 fever | 0 | 0
  Related fever | 1 | 0

4. Primary Outcome: Duration of Solicited General Symptoms
Description: Duration was expressed as median number of days any symptom persisted. Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any: occurrence of any general symptom regardless of their intensity grade or relationship to vaccination.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on those subjects who reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 8 | 5
Days
  Arthralgia (N= 8; 5) | 2.0 [1.0 to 5.0] | 3.0 [1.0 to 7.0]
  Fatigue (N= 8; 3) | 2.5 [1.0 to 6.0] | 1.0 [1.0 to 2.0]
  Headache (N= 8; 3) | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Myalgia (N= 8; 1) | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 1.0]
  Nausea (N= 3; 1) | 4.0 [2.0 to 4.0] | 2.0 [2.0 to 2.0]
  Shivering (N= 6; 3) | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fever (N= 1; 0) | NA [NA to NA] — Information on duration of fever was missing from this subject's symptom sheet. | NA [NA to NA] — None of the subjects in this group reported fever.

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any: occurrence of any unsolicited AE regardless of their intensity grade or relationship to vaccination. Grade 3: unsolicited AE that prevented normal everyday activities. Related: unsolicited AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 21-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 33 | 35
Subjects
  Any AEs | 5 | 7
  Grade 3 AEs | 1 | 0
  Related AEs | 1 | 2

6. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: Medically Significant Conditions (MSCs) included all unsolicited adverse events that resulted in a medically attended visit. Any: occurrence of any MSC regardless of their intensity grade or relationship to vaccination. Grade 3: MSC that prevented normal everyday activities. Related: MSC assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 21-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 33 | 35
Subjects
  Any MSCs | 2 | 4
  Grade 3 MSCs | 1 | 0
  Related MSCs | 0 | 0

7. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any: occurrence of any SAE regardless of their relationship to vaccination. Related: SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the entire study (up to Day 21)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 33 | 35
Subjects
  Any SAEs | 0 | 0
  Related SAEs | 0 | 0

8. Secondary Outcome: Serum Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Vaccine Strains
Description: Titers were expressed as Geometric Mean Titers. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity including all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 32 | 35
Titer
  A/Solomon Islands [Day 0] | 12.7 [8.8 to 18.2] | 9.0 [6.4 to 12.5]
  A/Solomon Islands [Day 21] | 63.0 [41.5 to 95.7] | 42.4 [28.3 to 63.5]
  A/Wisconsin [Day 0] | 100.3 [67.2 to 149.7] | 83.1 [63.1 to 109.5]
  A/Wisconsin [Day 21] | 252.2 [195.8 to 324.7] | 158.4 [114.1 to 219.7]
  B/Malaysia [Day 0] | 55.8 [37.4 to 83.3] | 61.2 [44.2 to 84.6]
  B/Malaysia [Day 21] | 126.1 [90.2 to 176.3] | 99.4 [74.2 to 133.3]

9. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against Each of the Three Vaccine Strains
Description: A seropositive subject was defined as a subject with a serum HI titer greater than or equal to 1:10. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 32 | 35
Subjects
  A/Solomon Islands [Day 0] | 18 | 15
  A/Solomon Islands [Day 21] | 29 | 32
  A/Wisconsin [Day 0] | 30 | 35
  A/Wisconsin [Day 21] | 32 | 35
  B/Malaysia [Day 0] | 31 | 34
  B/Malaysia [Day 21] | 32 | 35

10. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Each of the Three Vaccine Strains
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below1:10 and a post-vaccination titer greater than or equal to1:40 or a pre-vaccination titer greater than or equal to1:10 and at least a four-fold increase in post-vaccination titer. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 32 | 35
Subjects
  A/Solomon Islands | 20 | 17
  A/Wisconsin | 9 | 7
  B/Malaysia | 8 | 3

11. Secondary Outcome: Seroconversion Factors (SCFs) for HI Antibodies Against Each of the Three Vaccine Strains
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 32 | 35
fold increase
  A/Solomon Islands | 5.0 [3.3 to 7.5] | 4.7 [3.2 to 7.0]
  A/Wisconsin | 2.5 [2.0 to 3.1] | 1.9 [1.6 to 2.3]
  B/Malaysia | 2.3 [1.8 to 2.9] | 1.6 [1.4 to 1.9]

12. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against Each of the Three Vaccine Strains
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 32 | 35
Subjects
  A/Solomon Islands [Day 0] | 9 | 3
  A/Solomon Islands [Day 21] | 27 | 22
  A/Wisconsin [Day 0] | 29 | 31
  A/Wisconsin [Day 21] | 32 | 35
  B/Malaysia [Day 0] | 20 | 29
  B/Malaysia [Day 21] | 31 | 34

13. Secondary Outcome: Number of Cytokine-positive Cluster of Differentiation 4 (CD4) T Lymphocytes Per Million T Lymphocytes for Each of the Three Vaccine Strains
Description: Results are presented as geometric mean number of specific influenza CD4 T lymphocytes per million T lymphocytes. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia. Results are given for All doubles (i.e. CD4 T lymphocytes expressing at least 2 different cytokines [Cluster of Differentiation 40L (CD40L), Interleukin-2 (IL-2), Tumor Necrosis Factor alpha (TNF-α), Interferon gamma (IFN-γ)]) and for CD4 T lymphocytes expressing one particular cytokine (CD40L, IL-2, TNF-α, or IFN-γ) and least one other.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 30 | 32
Cells per million
  All Doubles A/Solomon Islands [Day 0] (N= 30; 32) | 611.15 (487.68) | 353.41 (289.83)
  All Doubles A/Solomon Islands [Day 21] (N= 25; 31) | 761.22 (783.59) | 285.45 (288.42)
  All Doubles A/Wisconsin [Day 0] (N= 30; 32) | 877.26 (529.44) | 476.38 (438.45)
  All Doubles A/Wisconsin [Day 21] (N= 25; 31) | 830.38 (652.85) | 357.12 (376.31)
  All Doubles B/Malaysia [Day 0] (N= 30; 32) | 643.26 (382.49) | 391.89 (285.28)
  All Doubles B/Malaysia [Day 21] (N= 25; 31) | 657.31 (542.67) | 200.13 (370.22)
  All Doubles Pooled Strains [Day 0] (N= 30; 32) | 1401.41 (671.68) | 767.10 (490.04)
  All Doubles Pooled Strains [Day 21] (N= 25; 31) | 1227.87 (1013.31) | 545.68 (480.37)
  CD40L A/Solomon Islands [Day 0] (N= 30; 32) | 606.58 (484.99) | 341.61 (291.23)
  CD40L A/Solomon Islands [Day 21] (N= 25; 31) | 758.40 (773.73) | 279.59 (284.97)
  CD40L A/Wisconsin [Day 0] (N= 30; 32) | 871.43 (512.44) | 472.33 (427.69)
  CD40L A/Wisconsin [Day 21] (N= 25; 31) | 829.38 (648.50) | 353.78 (377.73)
  CD40L B/Malaysia [Day 0] (N= 30; 32) | 640.49 (370.62) | 387.23 (280.03)
  CD40L B/Malaysia [Day 21] (N= 25; 31) | 648.93 (535.97) | 188.93 (361.66)
  CD40L Pooled Strains [Day 0] (N= 30; 32) | 1388.14 (661.04) | 757.53 (489.79)
  CD40L Pooled Strains [Day 21] (N= 25; 31) | 1209.75 (996.45) | 539.55 (476.23)
  IFN-γ A/Solomon Islands [Day 0] (N= 30; 32) | 393.40 (328.18) | 180.69 (182.12)
  IFN-γ A/Solomon Islands [Day 21] (N= 25; 31) | 411.23 (509.98) | 150.29 (185.78)
  IFN-γ A/Wisconsin [Day 0] (N= 30; 32) | 477.81 (299.82) | 232.70 (278.10)
  IFN-γ A/Wisconsin [Day 21] (N= 25; 31) | 357.56 (423.90) | 212.25 (191.16)
  IFN-γ B/Malaysia [Day 0] (N= 30; 32) | 405.44 (279.02) | 175.13 (210.56)
  IFN-γ B/Malaysia [Day 21] (N= 25; 31) | 442.51 (384.08) | 174.94 (229.30)
  IFN-γ Pooled Strains [Day 0] (N= 30; 32) | 824.34 (491.16) | 436.69 (307.38)
  IFN-γ Pooled Strains [Day 21] (N= 25; 31) | 840.65 (671.16) | 343.86 (315.56)
  IL-2 A/Solomon Islands [Day 0] (N= 30; 32) | 550.06 (433.42) | 321.49 (258.81)
  IL-2 A/Solomon Islands [Day 21] (N= 25; 31) | 635.35 (631.73) | 241.86 (225.01)
  IL-2 A/Wisconsin [Day 0] (N= 30; 32) | 738.42 (509.02) | 407.21 (381.85)
  IL-2 A/Wisconsin [Day 21] (N= 25; 31) | 682.25 (547.67) | 259.27 (313.49)
  IL-2 B/Malaysia [Day 0] (N= 30; 32) | 562.01 (340.18) | 377.10 (257.06)
  IL-2 B/Malaysia [Day 21] (N= 25; 31) | 577.43 (470.86) | 194.20 (319.95)
  IL-2 Pooled Strains [Day 0] (N= 30; 32) | 1192.89 (595.71) | 720.90 (421.55)
  IL-2 Pooled Strains [Day 21] (N= 25; 31) | 977.48 (819.44) | 463.25 (390.68)
  TNF-α A/Solomon Islands [Day 0] (N= 30; 32) | 270.39 (328.20) | 194.00 (169.53)
  TNF-α A/Solomon Islands [Day 21] (N= 25; 31) | 371.92 (409.87) | 129.21 (163.10)
  TNF-α A/Wisconsin [Day 0] (N= 30; 32) | 584.58 (352.86) | 334.97 (281.45)
  TNF-α A/Wisconsin [Day 21] (N= 25; 31) | 432.47 (428.19) | 271.33 (204.03)
  TNF-α B/Malaysia [Day 0] (N= 30; 32) | 278.06 (239.29) | 140.68 (165.67)
  TNF-α B/Malaysia [Day 21] (N= 25; 31) | 299.35 (322.28) | 102.33 (205.58)
  TNF-α Pooled Strains [Day 0] (N= 30; 32) | 794.15 (504.33) | 496.30 (298.79)
  TNF-α Pooled Strains [Day 21] (N= 25; 31) | 674.35 (584.50) | 251.59 (290.29)

14. Secondary Outcome: Number of Cytokine-positive Cluster of Differentiation 8 (CD8) T Lymphocytes Per Million T Lymphocytes for Each of the Three Vaccine Strains
Description: Results are presented as geometric mean number of specific influenza CD8 T lymphocytes per million T lymphocytes. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia. Results are given for All doubles (i.e. CD8 T lymphocytes expressing at least 2 different cytokines [Cluster of Differentiation 40L (CD40L), Interleukin-2 (IL-2), Tumor Necrosis Factor alpha (TNF-α), Interferon gamma (IFN-γ)]) and for CD8 T lymphocytes expressing one particular cytokine (CD40L, IL-2, TNF-α, or IFN-γ) and least one other.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Number analyzed (Participants) | 30 | 32
Cells per million
  All Doubles A/Solomon Islands [Day 0] (N= 30; 32) | 2.50 (54.81) | 3.01 (124.67)
  All Doubles A/Solomon Islands [Day 21] (N= 25; 31) | 6.18 (80.49) | 3.81 (52.84)
  All Doubles A/Wisconsin [Day 0] (N= 29; 32) | 5.48 (87.38) | 1.55 (40.24)
  All Doubles A/Wisconsin [Day 21] (N= 25; 31) | 3.11 (95.32) | 2.49 (55.29)
  All Doubles B/Malaysia [Day 0] (N= 29; 32) | 6.20 (90.23) | 2.51 (63.21)
  All Doubles B/Malaysia [Day 21] (N= 25; 31) | 3.26 (186.70) | 4.59 (70.75)
  All Doubles Pooled Strains [Day 0] (N= 29; 32) | 8.67 (123.74) | 4.43 (75.73)
  All Doubles Pooled Strains [Day 21] (N= 24; 31) | 10.96 (135.32) | 4.16 (98.01)
  CD40L A/Solomon Islands [Day 0] (N= 30; 32) | 2.05 (27.92) | 2.38 (57.63)
  CD40L A/Solomon Islands [Day 21] (N= 25; 31) | 5.00 (52.91) | 3.17 (44.66)
  CD40L A/Wisconsin [Day 0] (N= 29; 32) | 4.28 (60.42) | 1.55 (40.24)
  CD40L A/Wisconsin [Day 21] (N= 25; 31) | 2.14 (51.75) | 1.83 (41.14)
  CD40L B/Malaysia [Day 0] (N= 29; 32) | 6.59 (77.30) | 2.03 (45.49)
  CD40L B/Malaysia [Day 21] (N= 25; 31) | 3.08 (75.58) | 3.67 (64.11)
  CD40L Pooled Strains [Day 0] (N= 29; 32) | 6.61 (69.93) | 3.65 (58.75)
  CD40L Pooled Strains [Day 21] (N= 24; 31) | 6.37 (88.95) | 2.91 (87.43)
  IFN-γ A/Solomon Islands [Day 0] (N= 30; 32) | 1.77 (25.17) | 1.60 (123.31)
  IFN-γ A/Solomon Islands [Day 21] (N= 25; 31) | 1.40 (18.00) | 1.73 (23.95)
  IFN-γ A/Wisconsin [Day 0] (N= 29; 32) | 1.96 (58.89) | 1.52 (26.15)
  IFN-γ A/Wisconsin [Day 21] (N= 25; 31) | 1.41 (19.53) | 1.78 (33.55)
  IFN-γ B/Malaysia [Day 0] (N= 29; 32) | 3.18 (60.84) | 2.34 (63.80)
  IFN-γ B/Malaysia [Day 21] (N= 25; 31) | 1.92 (127.13) | 1.52 (22.73)
  IFN-γ Pooled Strains [Day 0] (N= 29; 32) | 2.39 (93.19) | 1.53 (30.78)
  IFN-γ Pooled Strains [Day 21] (N= 24; 31) | 3.24 (61.69) | 1.84 (39.83)
  IL-2 A/Solomon Islands [Day 0] (N= 30; 32) | 2.49 (54.69) | 2.46 (66.32)
  IL-2 A/Solomon Islands [Day 21] (N= 25; 31) | 4.39 (76.84) | 3.38 (48.89)
  IL-2 A/Wisconsin [Day 0] (N= 29; 32) | 5.27 (69.84) | 1.76 (41.38)
  IL-2 A/Wisconsin [Day 21] (N= 25; 31) | 2.63 (95.37) | 1.82 (38.90)
  IL-2 B/Malaysia [Day 0] (N= 29; 32) | 4.86 (77.20) | 1.78 (44.85)
  IL-2 B/Malaysia [Day 21] (N= 25; 31) | 2.60 (75.43) | 3.72 (63.72)
  IL-2 Pooled Strains [Day 0] (N= 29; 32) | 7.44 (95.70) | 6.54 (69.82)
  IL-2 Pooled Strains [Day 21] (N= 24; 31) | 6.63 (107.41) | 3.39 (91.57)
  TNF-α A/Solomon Islands [Day 0] (N= 30; 32) | 1.58 (23.46) | 2.77 (101.63)
  TNF-α A/Solomon Islands [Day 21] (N= 25; 31) | 2.47 (55.20) | 2.67 (36.03)
  TNF-α A/Wisconsin [Day 0] (N= 29; 32) | 2.36 (69.91) | 1.31 (18.78)
  TNF-α A/Wisconsin [Day 21] (N= 25; 31) | 2.08 (53.64) | 2.03 (32.51)
  TNF-α B/Malaysia [Day 0] (N= 29; 32) | 3.09 (61.50) | 3.29 (77.18)
  TNF-α B/Malaysia [Day 21] (N= 25; 31) | 1.92 (127.13) | 1.83 (34.42)
  TNF-α Pooled Strains [Day 0] (N= 29; 32) | 2.37 (82.35) | 1.59 (50.66)
  TNF-α Pooled Strains [Day 21] (N= 24; 31) | 4.12 (88.07) | 2.38 (37.12)

ADVERSE EVENTS:
Time Frame: Events collected by systematic assessment: 7-day follow-up period after vaccination. Events collected by non-systematic assessment: 21-day follow-up period after vaccination.
Arm/Group | FluAS25 (GSK576389A) Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 24/33 | 17/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FluAS25 (GSK576389A) Group (N=33) | Fluarix Group (N=35)
Pain (General disorders) | 17 | 7
Swelling (General disorders) | 2 | 2
Redness (General disorders) | 10 | 4
Arthralgia (General disorders) | 8 | 5
Fatigue (General disorders) | 8 | 3
Headache (General disorders) | 8 | 3
Myalgia (General disorders) | 8 | 1
Nausea (General disorders) | 3 | 1
Shivering (General disorders) | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Injection site pruritus (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.